CLINICAL TRIAL: NCT03113656
Title: The Use of Weighted Blankets in the Care of Infants With Neonatal Abstinence Syndrome (NAS)
Brief Title: Weighted Blankets With Infants With NAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Principal Investigator, Rachel Baker, Nurse Researcher, TriHealth Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 17-008
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weighted Blanket First (Experimental): This group will receive the Weighted Blanket first and then the Non-weighted blanket
  Interventions: Other: Weighted Blanket; Other: Non-Weighted Blanket
- Non-weighted Blanket First (Experimental): This group will receive the Non-weighted Blanket first and then the Weighted blanket
  Interventions: Other: Weighted Blanket; Other: Non-Weighted Blanket

INTERVENTIONS:
Other: Weighted Blanket — Weighted blanket placed on infant for 30 minutes
Other: Non-Weighted Blanket — Non-Weighted blanket placed on infant for 30 minutes

SUMMARY:
Infants with neonatal abstinence syndrome (NAS) who are cared for in a Neonatal Intensive Care Unit (NICU) often display symptoms including hyperactivity, irritability, jitteriness, poor feeding, and poor sleep patterns. The recommended first line of treatment to relieve these symptoms involves nonpharmacological interventions. The purpose of the current pilot study is to provide preliminary data to assist in the design of a larger scale study to examine one nonpharmacological intervention, weighted blankets. The pilot study will assess the feasibility of a cross-over randomized controlled design to study the impact of a weighted blanket on infants' symptoms of NAS.

The aims of the study are:

Aim1: To determine the feasibility of recruiting patients for a study evaluating the use of weighted blankets in the care of infants with NAS Aim 2: To determine the feasibility and safety of the study procedures Aim 3: To examine whether there is clinical benefit to using weighted blankets for the treatment of symptoms in infants with NAS.

After informed consent is obtained, infants will be randomized to have either a weighted blanket or a non-weighted blanket placed on them first. A cross-over design will be used so all infants will experience both the non-weighted and weighted blankets. Thirty minutes before each feeding, baseline vital signs and Finnegan score will be obtained. Then, a blanket (weighted or non-weighted) will be placed on the infant for 30 minutes. Infants will be directly monitored and on heart rate/respiratory rate monitors while the blanket is applied. Vital signs and Finnegan scores will be obtained at the end of 30 minutes of blanket placement, infants will be fed, and vital signs and Finnegan scores will be obtained again 30 minutes after the blanket was removed. Descriptive statistics will be used to determine the enrollment rate and feasibility of the protocol. Nonparametric statistics will be used to compare total Finnegan scores for infants with the weighted blanket applied compared to infants with a non-weighted blanket applied. Changes in Finnegan scores will be examined to estimate an effect size to use in a power analysis for a future larger effectiveness study.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the NICU
* Gestational age > 37 weeks
* Positive maternal drug screen at delivery

Exclusion Criteria:

* Clinical staff does not give permission to enroll the patient
* Had intrauterine growth restriction (IUGR)
* Has any medical diagnosis in addition to NAS diagnosis
* Has a weight below the 10th percentile

Min Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Weighted Blanket First | Non-weighted Blanket First
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weighted Blanket First | Non-weighted Blanket First | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: days] | 6.89 (8.24) | 4.00 (3.06) | 5.63 (6.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 5 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Finnegan Score
Description: Finnegan scale measures signs of neonatal drug withdrawal syndrome. It provides a summative score obtained from the assessment of 21 items related to neonatal withdrawal. The total score ranges from 0 to 43 with a higher score indicating more severe symptoms. Values above 8 have been described as being indicative of neonatal abstinence syndrome.
Time Frame: baseline and 30 minutes
Population: Reporting Arms/Groups "per intervention"
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention: Weighted Blanket: Weighted blanket placed on infant for 30 minutes
- Control: Non-Weighted Blanket: Non-Weighted blanket placed on infant for 30 minutes
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 16
score on a scale | -1.5167 (2.251) | -0.2549 (1.787)

ADVERSE EVENTS:
Time Frame: During entire hospitalization (ranged from 1 day to 15 days)
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT03113656/Prot_SAP_000.pdf